CLINICAL TRIAL: NCT03064152
Title: Rotational Thromboelastometry for the Transfusion Management of Postpartum Hemorrhage After Vaginal or Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment, outcome measures collected but actual enrollment is below target enrollment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michaela Kristina Farber, MD, Principle Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001800
Record Dates: First submitted 2017-02-17; First posted 2017-02-24 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Patients who experience postpartum hemorrhage will receive standard of care for labor and delivery, cesarean delivery, and postpartum care. Transfusion will be based on standard of care utilizing clinical criteria of hemodynamics (noninvasive blood pressure, heart rate, arterial line if deemed clinically useful) and coagulation labs (PT, activated partial thromboplastin time (aPTT), fibrinogen, complete blood count). In addition to standard of care, additional ROTEM blood assays will be performed at any time routine coagulation labs are sent. Providers in the control group will be blinded to ROTEM results.
- ROTEM (Experimental): Patients will receive standard of care for labor and delivery, cesarean delivery, and postpartum care. Transfusion will be based on standard of care utilizing clinical criteria of hemodynamics (noninvasive blood pressure, heart rate, arterial line if deemed clinically useful) and coagulation labs (PT, aPTT, fibrinogen, complete blood count). In addition to standard of care, additional ROTEM blood assays will be performed at any time routine coagulation labs are sent. Providers in the ROTEM group will receive real-time ROTEM results and a previously validated ROTEM-based transfusion algorithm for PPH.
  Interventions: Device: Rotational Thromboelastometry

INTERVENTIONS:
Device: Rotational Thromboelastometry — ROTEM is a point-of-care coagulation assay.
  Other Names: ROTEM
  Arms: ROTEM

SUMMARY:
The aim of this study is to evaluate the impact of a rotational thromboelastometry (ROTEM®)-based transfusion protocol during postpartum hemorrhage (PPH) after vaginal or cesarean delivery. Maternal transfusion requirement, quantitative blood loss (QBL), need for intensive care unit (ICU) admission, and length of hospital stay will be evaluated. The utilization of ROTEM® for transfusion management will identify patients who develop early coagulation changes such as hypofibrinogenemia or disseminated intravascular coagulation. Our hypothesis is that earlier identification and directed therapy of such coagulation changes will lower overall transfusion requirement (packed red blood cells, fresh frozen plasma, fibrinogen concentrate, cryoprecipitate, or other product), reduce the need for ICU admission, and shorten length of hospital stay. A cost analysis will be performed.

DETAILED DESCRIPTION:
Postpartum hemorrhage is increasing in incidence in the United States, renewing interest in targeted approaches to transfusion during cesarean delivery. ROTEM-based transfusion for PPH has been advocated as a mechanism to lower overall requirement of blood components transfused and lower the incidence of transfusion-associated pulmonary morbidity in a small study of women undergoing cesarean delivery. However, larger-scale randomized evaluation of this transfusion approach is warranted for women who experience hemorrhage after vaginal or cesarean delivery. A lower serum fibrinogen level (< 200 mg/dL) at the onset of PPH has a positive predictive value of 100% for progression to severe PPH. However, serum fibrinogen testing has a turnaround time of one hour and is therefore not useful for acute management of PPH. ROTEM provides point-of-care results that have been validated as surrogate markers for serum fibrinogen, within 10 minutes. However, whether ROTEM data alters empiric management of acute PPH is unknown. A comparison of transfusion management decisions and costs incurred for transfused products and transfusion-related morbidity (duration of hospitalization, intensive care unit, respiratory complications) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) II or III health status (minimal to no systemic disease), age between 18 and 50 yrs, singleton pregnancies admitted for labor and delivery anticipated or actual PPH, or anticipated transfusion of blood products. This will be defined by one or more of the following eligibility criteria:

  1. Cesarean delivery with moderate or high risk for PPH (see below).
  2. Cesarean delivery with acute PPH of > 1000 mL and blood products ordered from the blood bank.
  3. Vaginal delivery with acute PPH of > 500 mL and blood products ordered from the blood bank.

For criterion #1, moderate risk for PPH is defined by one or more of the following features:

* prior cesarean delivery in labor
* prior cesarean delivery with known adhesive disease of the placenta
* multiple gestation
* >4 previous vaginal births
* chorioamnionitis with maternal temperature > 101 degrees Fahrenheit
* history of previous PPH
* large uterine fibroids (> 5 cm)
* second stage of labor (10cm cervical dilation to delivery) > 3 hours

High risk for postpartum hemorrhage is defined by one or more of the following features:

* suspected placenta accreta by pre-delivery ultrasound findings
* placenta previa (current or resolved within 4 weeks of delivery) or low-lying placenta
* active bleeding on admission prior to delivery

Exclusion Criteria:

* known coagulation defect prior to delivery including inherited (hemophilia A, von Willebrand disease, thrombocytopenia, other) or iatrogenic causes (anticoagulation therapy), refusal to accept blood transfusion (Jehovah's Witness, other).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michaela K Farber, MD MS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | ROTEM
Started | 26 | 23
Completed | 26 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: same as Participant Flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | ROTEM | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (5.2) | 36.0 (5.2) | 36.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 26 | 23 | 49
  Sex: Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 22 | 46
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 17 | 14 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
weight (kg) [Mean (Standard Deviation); unit: kg] | 87 (18.7) | 82.5 (15.7) | 85 (16.5)
height [Mean (Standard Deviation); unit: inches] | 64.8 (3.4) | 64.4 (2.1) | 64.5 (2.5)
body mass index ( kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 33.7 (9.4) | 30.7 (6.0) | 32.0 (7.0)
gestational age [Mean (Standard Deviation); unit: weeks] | 36.6 (1.9) | 36.0 (2.3) | 36.4 (2.0)
gravidity [Median (Inter-Quartile Range); unit: pregnancies] | 3 [2 to 4] | 4 [2 to 5] | 3 [2 to 5]
parity [Median (Inter-Quartile Range); unit: deliveries] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
twin gestation (n) [Count of Participants; unit: Participants] | 3 | 3 | 6
anesthesia type [Number; unit: participants]
  combined spinal epidural | 14 | 15 | 29
  epidural | 4 | 3 | 7
  general | 2 | 0 | 2
  spinal | 6 | 5 | 11
delivery type [Number; unit: participants]
  scheduled cesarean delivery | 20 | 19 | 39
  unscheduled cesarean delivery | 5 | 3 | 8
  vaginal delivery | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Total Blood Products Transfused Within 48h of Onset of PPH
Description: Total number of packed red blood cells (PRBCs), fresh frozen plasma (FFP), platelets, cryoprecipitate, cell salvage units within 48h of onset of PPH
Time Frame: t0 = diagnosis of PPH by criteria defined; t final = 48h after onset of PPH.
Measure: Median (Inter-Quartile Range); unit: blood products
Arm/Group | Control | ROTEM
Number analyzed (Participants) | 26 | 23
blood products | 2 [1 to 5.1] | 1.4 [0 to 7]

2. Secondary Outcome: Blood Loss
Description: Visual estimate in suction canister and sponges, or quantitative blood loss
Time Frame: From the onset of PPH through 4 hours from leaving the operating room or within 4 hours from the last blood transfusion, whichever occurs later and on average 5 hours.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Control | ROTEM
Number analyzed (Participants) | 26 | 23
mL | 2000 [1500 to 2600] | 2100 [1800 to 2844]

3. Secondary Outcome: Number of Participants With Admission to the Intensive Care Unit
Description: Number of participants needing admission to the intensive care unit within 2 weeks of delivery
Time Frame: within 2 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | ROTEM
Number analyzed (Participants) | 26 | 23
Participants | 1 | 2

4. Secondary Outcome: Number of Participants Who Required a Hysterectomy
Description: Number of participants who required a hysterectomy to control postpartum hemorrhage.
Time Frame: within 2 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | ROTEM
Number analyzed (Participants) | 26 | 23
Participants | 14 | 13

5. Secondary Outcome: Number of Participants Who Experienced Maternal Mortality
Description: Number of participants who experienced maternal death after delivery.
Time Frame: within 2 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | ROTEM
Number analyzed (Participants) | 26 | 23
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Each enrolled participant was directly involved in the study for approximately 3-5 hours for the duration of their time in the operating room, until the end of follow-up, up to 2 weeks postpartum.
Description: As described by clinicaltrials.gov.
Arm/Group | Control | ROTEM
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT03064152/Prot_SAP_000.pdf